CLINICAL TRIAL: NCT03462082
Title: A Single-center, Randomized, Double-blinded, Double-crossover Trial of Asymmetric Subthalamic Deep Brain Stimulation for Axial Motor Dysfunction in Parkinson's Disease
Brief Title: Asymmetric Subthalamic Deep Brain Stimulation for Axial Motor Dysfunction in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Alfonso Fasano, Professor, University of Toronto
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-5785
Record Dates: First submitted 2018-03-05; First posted 2018-03-12 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; axial motor dysfunction; asymmetric neuromodulation; subthalamic nucleus deep brain stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Baseline STN-DBS (No Intervention): Maintenance of baseline bilateral STN-DBS settings.
- Asymmetric STN-DBS 1 (Experimental): Unilateral 50% reduction of voltage (e.g. right side)
  Interventions: Other: Asymmetric STN-DBS
- Asymmetric STN-DBS 2 (Experimental): Unilateral 50% reduction of voltage (e.g. left side)
  Interventions: Other: Asymmetric STN-DBS

INTERVENTIONS:
Other: Asymmetric STN-DBS — Asymmetric deep brain stimulation
  Arms: Asymmetric STN-DBS 1; Asymmetric STN-DBS 2

SUMMARY:
This single-center, randomized, quadruple-blinded, double-crossover comparative efficacy trial will study the effects of unilateral 50% voltage reduction in axial motor dysfunction for patients with Parkinson's disease that develop treatment-resistant postural stability gait dysfunction after bilateral subthalamic nucleus deep brain stimulation surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease (PD) (previously diagnosed according to the UK brain bank criteria) who develop treatment-resistant postural instability gait dysfunction (PIGD) more than 6 months but less than 5 years after bilateral subthalamic nucleus deep brain stimulation (STN-DBS).
* Treatment-resistant PIGD will be defined as freezing of gait and UPDRS or MDS-UPDRS PIGD subscales of more than 6 points despite optimization of medications and bilateral STN-DBS programming.

Exclusion Criteria:

* Treatment-resistant PIGD less than 6 months or more than 5 years after STN-DBS surgery.
* PIGD responsive to optimization of medications and/or bilateral STN-DBS programming.
* Cognitive impairment or psychiatric comorbidities (including substance abuse) that would interfere with the informed consent process, study adherence or outcome assessments.
* Advanced PD or any other neurological, cardiovascular or musculoskeletal co-morbidities that would preclude or require assistance to complete the 10-meter walking test.
* Patients not able to comply with 4-week interval evaluations following their potential enrollment due to personal reasons.
* Serious illness (requiring systemic treatment and/or hospitalization) until subject either completes therapy or is clinically-stable on therapy, in the opinion of the site investigator, for at least 30 days prior to study entry.
* Inability or unwillingness of subject or legal guardian/representative to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-03-14 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Fasano, MD, PhD, Principal Investigator — University of Toronto
Locations (1):
- Movement disorders Centre, Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
To be shared as supplementary data upon publication of the results of the trial.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: To be shared as supplementary data upon publication of the results of the trial.

REFERENCES:
- [Background] Fasano A, Herzog J, Seifert E, Stolze H, Falk D, Reese R, Volkmann J, Deuschl G. Modulation of gait coordination by subthalamic stimulation improves freezing of gait. Mov Disord. 2011 Apr;26(5):844-51. doi: 10.1002/mds.23583. Epub 2011 Mar 2. PMID 21370271
- [Background] Lizarraga KJ, Jagid JR, Luca CC. Comparative effects of unilateral and bilateral subthalamic nucleus deep brain stimulation on gait kinematics in Parkinson's disease: a randomized, blinded study. J Neurol. 2016 Aug;263(8):1652-6. doi: 10.1007/s00415-016-8191-3. Epub 2016 Jun 8. PMID 27278062
- [Background] Lizarraga KJ, Luca CC, De Salles A, Gorgulho A, Lang AE, Fasano A. Asymmetric neuromodulation of motor circuits in Parkinson's disease: The role of subthalamic deep brain stimulation. Surg Neurol Int. 2017 Oct 24;8:261. doi: 10.4103/sni.sni_292_17. eCollection 2017. PMID 29184712
- [Derived] Lizarraga KJ, Gnanamanogaran B, Al-Ozzi TM, Cohn M, Tomlinson G, Boutet A, Elias GJB, Germann J, Soh D, Kalia SK, Hodaie M, Munhoz RP, Marras C, Hutchison WD, Lozano AM, Lang AE, Fasano A. Lateralized Subthalamic Stimulation for Axial Dysfunction in Parkinson's Disease: A Randomized Trial. Mov Disord. 2022 May;37(5):1079-1087. doi: 10.1002/mds.28953. Epub 2022 Feb 13. PMID 35156734

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 patients with Parkinson's disease (PD) who developed postural instability gait dysfunction (PIGD) after bilateral subthalamic (STN) deep brain stimulation (DBS) were screened for eligibility between January 22, 2018 and January 29, 2019 at the DBS clinic of the Movement Disorders Center at the University of Toronto in Toronto, Ontario, Canada.
Pre-assignment Details: 22 of 38 patients were enrolled. Of the 16 patients not enrolled, 9 did not meet inclusion criteria and 7 declined to participate.
  There were no significant events between enrollment and randomization.
  The first study participant was enrolled on March 14, 2018. The last study participant was enrolled on January 29, 2019.
Groups:
- Bilateral DBS Then Asymmetric DBS 1 Then Asymmetric DBS 2: Baseline bilateral STN-DBS for 3 to 4 weeks, followed by asymmetric STN-DBS 1 (right STN-DBS amplitude reduced by 50%) for 3 to 4 weeks, followed by asymmetric STN-DBS 2 (left STN-DBS amplitude reduced by 50%) for 3 to 4 weeks.
- Bilateral DBS Then Asymmetric DBS 2 Then Asymmetric DBS 1: Baseline bilateral STN-DBS for 3 to 4 weeks, followed by asymmetric STN-DBS 2 (left STN-DBS amplitude reduced by 50%) for 3 to 4 weeks, followed by asymmetric STN-DBS 1 (right STN-DBS amplitude reduced by 50%) for 3 to 4 weeks.
- Asymmetric DBS 1 Then Bilateral DBS Then Asymmetric DBS 2: Asymmetric STN-DBS 1 (right STN amplitude reduced by 50%) for 3 to 4 weeks, followed by baseline bilateral STN-DBS for 3 to 4 weeks, followed by asymmetric STN-DBS 2 (left STN-DBS amplitude reduced by 50%) for 3 to 4 weeks.
- Asymmetric DBS 1 Then Asymmetric DBS 2 Then Bilateral DBS: Asymmetric STN-DBS 1 (right STN-DBS amplitude reduced by 50%) for 3 to 4 weeks, followed by asymmetric STN-DBS 2 (left STN-DBS amplitude reduced by 50%) for 3 to 4 weeks, followed by baseline bilateral STN-DBS for 3 to 4 weeks.
- Asymmetric DBS 2 Then Bilateral DBS Then Asymmetric DBS 1: Asymmetric STN-DBS 2 (left STN-DBS amplitude reduced by 50%) for 3 to 4 weeks, followed by baseline bilateral STN-DBS for 3 to 4 weeks, followed by asymmetric STN-DBS 1 (right STN-DBS amplitude reduced by 50%) for 3 to 4 weeks.
- Asymmetric DBS 2 Then Asymmetric DBS 1 Then Bilateral DBS: Asymmetric STN-DBS 2 (left STN-DBS amplitude reduced by 50%) for 3 to 4 weeks, followed by asymmetric STN-DBS 1 (right STN-DBS amplitude reduced by 50%) for 3 to 4 weeks, followed by baseline bilateral STN-DBS for 3 to 4 weeks.
- Asymmetric DBS 1 (Open Label): After the Study Phase (Randomized, Blinded Period) was completed, patients were offered to participate in an Open Label Phase in which they would be switched for at least 12 weeks to either the Asymmetric DBS 1 or the Asymmetric DBS 2 condition if it was associated with axial symptom improvement when compared to their baseline bilateral DBS condition.
  Out of the 22 patients initially enrolled, 17 opted to participate. Out of the 17 patients that opted to participate, 7 were switched to the Asymmetric DBS 1 condition: 50% reduction of right STN-DBS amplitude (voltage)
- Asymmetric DBS 2 (Open Label): After the Study Phase (Randomized, Blinded Period) was completed, patients were offered to participate in an Open Label Phase in which they would be switched for at least 12 weeks to either the Asymmetric DBS 1 or the Asymmetric DBS 2 condition if it was associated with axial symptom improvement when compared to their baseline bilateral DBS condition.
  Out of the 22 patients initially enrolled, 17 opted to participate. Out of the 17 patients that opted to participate, 10 were switched to the Asymmetric DBS 2 condition: 50% reduction of left STN-DBS amplitude (voltage)
Period: Study Phase (Randomized, Blinded Period)
Arm/Group | Bilateral DBS Then Asymmetric DBS 1 Then Asymmetric DBS 2 | Bilateral DBS Then Asymmetric DBS 2 Then Asymmetric DBS 1 | Asymmetric DBS 1 Then Bilateral DBS Then Asymmetric DBS 2 | Asymmetric DBS 1 Then Asymmetric DBS 2 Then Bilateral DBS | Asymmetric DBS 2 Then Bilateral DBS Then Asymmetric DBS 1 | Asymmetric DBS 2 Then Asymmetric DBS 1 Then Bilateral DBS | Asymmetric DBS 1 (Open Label) | Asymmetric DBS 2 (Open Label)
Started | 3 | 4 | 4 | 3 | 3 | 5 | 0 | 0
Completed | 3 | 4 | 4 | 3 | 3 | 5 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open Label Phase
Arm/Group | Bilateral DBS Then Asymmetric DBS 1 Then Asymmetric DBS 2 | Bilateral DBS Then Asymmetric DBS 2 Then Asymmetric DBS 1 | Asymmetric DBS 1 Then Bilateral DBS Then Asymmetric DBS 2 | Asymmetric DBS 1 Then Asymmetric DBS 2 Then Bilateral DBS | Asymmetric DBS 2 Then Bilateral DBS Then Asymmetric DBS 1 | Asymmetric DBS 2 Then Asymmetric DBS 1 Then Bilateral DBS | Asymmetric DBS 1 (Open Label) | Asymmetric DBS 2 (Open Label)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Not completed — Symptom worsening (Treatment failure) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: Different arms/groups/sequences are combined because all 22 study participants received all treatments in the randomized/blinded phase of the study. The subsequent open label phase was optional and based on the results of the randomized/blinded phase.
Groups:
- All Study Participants: All Study Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 65.5 [51 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 22
Hand dominance [Median (Full Range); unit: units on a scale] — Laterality Index as measured by the Edinburgh inventory: Scale range is -100 (minimum) to 100 (maximum), -100 indicates complete left handedness and 100 indicates complete right handedness.
  units on a scale | 82.5 [-90 to 100]
Parkinson's disease duration [Median (Full Range); unit: years] | 17 [8.5 to 30.5]
Predominant motor symptom at onset [Count of Participants; unit: Participants]
  Tremor | 9
  Stiffness and/or Slowness | 13
More affected hemibody at onset [Count of Participants; unit: Participants]
  Right | 13
  Left | 8
  Both | 1
Indication for STN-DBS surgery [Count of Participants; unit: Participants]
  Medication-resistant tremor | 8
  Medication-resistant motor fluctuations | 14
Time since STN-DBS surgery [Median (Full Range); unit: months] | 51 [6 to 171]
Time between STN-DBS surgery and onset of axial dysfunction [Mean (Full Range); unit: months] | 14.5 [6 to 58]
More affected hemibody at enrollment [Count of Participants; unit: Participants]
  Right | 4
  Left | 4
  Both | 14
Levodopa equivalent daily dose [Median (Full Range); unit: mg/day] | 1037.5 [600 to 2263]
Baseline right STN-DBS type [Count of Participants; unit: Participants]
  Conventional monopolar | 1
  Low-frequency monopolar | 8
  High-frequency monopolar | 3
  Interleaving low-frequency monopolar | 4
  Double low-frequency monopolar | 1
  Interleaving low-frequency monopolar/double monop. | 1
  Conventional bipolar | 1
  Low-frequency bipolar | 2
  High-frequency bipolar | 0
  Interleaving conventional monopolar / bipolar | 1
Baseline right STN-DBS amplitude [Median (Full Range); unit: Volts] | 3.95 [1.85 to 7.1]
Baseline right STN-DBS frequency [Median (Full Range); unit: Hertz] | 80 [50 to 185]
Baseline right STN-DBS pulse width [Median (Full Range); unit: Microseconds] | 60 [60 to 60]
Baseline total electrical energy delivered (TEED) to the right STN [Median (Full Range); unit: Joules/second] — Formula:
  TEED = (Voltage)(Voltage)*(Pulse Width)*(Frequency) / (Impedance)
  Joules/second | 88.59 [19.88 to 240.06]
Baseline left STN-DBS type [Count of Participants; unit: Participants]
  Conventional monopolar | 0
  Low-frequency monopolar | 8
  High-frequency monopolar | 1
  Interleaving low-frequency monopolar | 4
  Double low-frequency monopolar | 0
  Interleaving low-frequency monopolar/double monop. | 1
  Conventional bipolar | 2
  Low-frequency bipolar | 3
  High-frequency bipolar | 2
  Interleaving conventional monopolar / bipolar | 1
Baseline left STN-DBS amplitude [Median (Full Range); unit: Volts] | 4.08 [2.2 to 7.1]
Baseline left STN-DBS frequency [Median (Full Range); unit: Hertz] | 80 [50 to 185]
Baseline left STN-DBS pulse width [Median (Full Range); unit: Microseconds] | 60 [60 to 60]
Baseline total electrical energy delivered (TEED) to the left STN [Median (Full Range); unit: Joules/second] — Formula:
  TEED = (Voltage)(Voltage)*(Pulse Width)*(Frequency) / (Impedance)
  Joules/second | 89.66 [29.75 to 399.6]
Gait velocity [Mean (Full Range); unit: m/s] — As measured during the 10-meter walk test. In this test, participants walk at their usual, regular pace over a total distance of 10 meters. The middle 6-meters (between the 2-meter and 8-meter marks) are timed to measure gait velocity during steady-state gait.
  m/s | 0.976 [0.272 to 1.322]
MDS-UPDRS (total) [Median (Full Range); unit: units on a scale] — The MDS-UPDRS (Movement Disorders Society Unified Parkinson's Disease Rating Scale) is a clinical and research tool to measure symptoms and signs of Parkinson's disease. It has 4 parts: Part I (non-motor experiences of daily living), Part II (motor experiences of daily living), Part III (motor examination) and Part IV (motor complications). The MDS-UPDRS has a total of 60 items, scored from 0-4 each. The minimum score is 0 and the maximum score is 240. Lower scores indicate better and higher scores indicate worse symptoms and signs of Parkinson's disease, respectively.
  units on a scale | 89 [62 to 151]
MDS-UPDRS (motor) [Median (Full Range); unit: units on a scale] — The MDS-UPDRS (motor) is Part III of the Movement Disorders Society Unified Parkinson's Disease Rating Scale. It is a clinical and research tool to measure motor signs of Parkinson's disease. Part III of the MDS-UPDRS has 28 items, scored from 0-4 each, so the minimum score is 0 and the maximum score is 112. Lower scores indicate better and higher scores indicate worse motor signs of Parkinson's disease, respectively.
  units on a scale | 45.5 [34 to 71]
MDS-UPDRS (axial motor) [Median (Full Range); unit: units on a scale] — The MDS-UPDRS (axial motor) is composed of items 3.1 to 3.3a and 3.9 to 3.13 of the Part III of the Movement Disorders Society Unified Parkinson's Disease Rating Scale. It is a clinical and research tool to measure axial motor signs of Parkinson's disease. MDS-UPDRS (axial motor) has 8 items, scored from 0-4 each, so the minimum score is 0 and the maximum score is 32. Lower scores indicate better and higher scores indicate worse axial motor signs of Parkinson's disease, respectively.
  units on a scale | 16.5 [9 to 27]
Mini-BESTest score [Median (Full Range); unit: units on a scale] — The Mini-BESTest is a shorter version of the BESTest (Balance Evaluation Systems Test). It is a clinical and research tool to measure balance control.
  The Mini-BESTest has 14 items, scored from 0-2 each, so the minimum score is 0 and the maximum score is 28. Lower scores indicate worse balance control and higher scores indicate better balance control.
  units on a scale | 15 [2 to 21]
UPDRS-PIGD score [Median (Full Range); unit: units on a scale] — The UPDRS-PIGD is the Postural Instability Gait Dysfunction (PIGD) sub-scale of the Unified Parkinson's Disease Rating Scale (UPDRS). It is a clinical and research tool to measure PIGD.
  The UPDRS-PIGD has 5 items, scored from 0-4 each, so the minimum score is 0 and the maximum score is 20. Lower scores indicate better PIGD and higher scores indicate worse PIGD.
  units on a scale | 11 [8 to 17]
Freezing of gait questionnaire [Median (Full Range); unit: units on a scale] — The Freezing of Gait Questionnaire is a clinical and research tool to measure freezing of gait. It has 6 items, scored from 0-4 each, so the minimum score is 0 and the maximum score is 24. Lower scores indicate better and higher scores indicate worse freezing of gait, respectively.
  units on a scale | 14.5 [7 to 23]
Summary index of the PDQ-39 [Median (Full Range); unit: units on a scale] — The 39-item Parkinson's Disease Quality of Life Questionnaire (PDQ-39) is a clinical and research tool to measure quality of life in Parkinson's disease. It has 39 questions, which patients score as never (0% of the time), occasionally (25% of the time), sometimes (50% of the time), often (75% of the time) or always (100% of the time). The PDQ-39 Total Score or Summary Index is the average of the 39 questions. The minimum score is 0% (never) and the maximum score is 100% (always). Lower scores indicate better quality of life and higher scores indicate worse quality of life.
  units on a scale | 31.54 [14.64 to 49.84]
Select cognitive tasks [Mean (Standard Deviation); unit: units on a scale] — Left brain cognitive function: Hopkins Verbal Learning Test-Revised: Total recall trials 1-3 (0-36), delayed recall (0-12); Phonemic Verbal Fluency (0-no max); Semantic Verbal Fluency (Animal cue) (0-no max); Letter 1-back and 2-back working memory tasks (0-100%). Right brain cognitive function: Brief Visual Memory Test-Revised: Total recall trials 1-3 (0-36), delayed recall (0-12); Computerized landmark line bisection (-10 to 10); Spatial 1-back and 2-back working memory tasks (0-100%). Ranges in parentheses. Line bisection: closer to 0 is more accurate. For the rest: higher values are better Population: Two patients could not complete cognitive tasks due to language barrier.
  units on a scale
    HopkinsVerbalLearningTest-Revised: RecallTrials1-3: number analyzed (Participants) | 20
    HopkinsVerbalLearningTest-Revised: RecallTrials1-3 | 21.75 (5.78)
    HopkinsVerbal LearningTest-Revised: Delayed Recall: number analyzed (Participants) | 20
    HopkinsVerbal LearningTest-Revised: Delayed Recall | 7.70 (2.56)
    Phonemic Verbal Fluency: number analyzed (Participants) | 20
    Phonemic Verbal Fluency | 31.50 (14.15)
    Semantic Verbal Fluency (Animal cue): number analyzed (Participants) | 20
    Semantic Verbal Fluency (Animal cue) | 16.80 (7.82)
    Letter 1-Back Working Memory Task: number analyzed (Participants) | 20
    Letter 1-Back Working Memory Task | 82.86 (18.51)
    Letter 2-Back Working Memory Task: number analyzed (Participants) | 20
    Letter 2-Back Working Memory Task | 55.11 (26.28)
    Brief Visual Memory Test-Revised: RecallTrials 1-3: number analyzed (Participants) | 20
    Brief Visual Memory Test-Revised: RecallTrials 1-3 | 12.75 (6.24)
    Brief Visual Memory Test-Revised: Delayed Recall: number analyzed (Participants) | 20
    Brief Visual Memory Test-Revised: Delayed Recall | 5.15 (3.38)
    Computerized landmark line bisection task: number analyzed (Participants) | 20
    Computerized landmark line bisection task | 0.08 (0.53)
    Spatial 1-Back Working Memory Task: number analyzed (Participants) | 20
    Spatial 1-Back Working Memory Task | 85.20 (23.22)
    Spatial 2-Back Working Memory Task: number analyzed (Participants) | 20
    Spatial 2-Back Working Memory Task | 57.81 (29.10)

OUTCOME MEASURES:

1. Primary Outcome: Change in Gait Velocity
Description: As measured during the 10-meter walk test. In this test, participants walk at their usual, regular pace over a total distance of 10 meters. The middle 6-meters (between the 2-meter and 8-meter marks) are timed to measure gait velocity during steady-state gait.
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: Bilateral (baseline) values are the average of the outcome measure data obtained during the 2 bilateral (baseline) conditions: 1) at enrollment before randomization and 2) after randomization. These average values are used to report the changes associated with the 2 asymmetric conditions.
Measure: Least Squares Mean (Standard Error); unit: m/s
Groups:
- Bilateral STN-DBS: Bilateral (baseline) STN-DBS settings
- Asymmetric STN-DBS 1: 50% reduction of right STN-DBS amplitude (voltage)
- Asymmetric STN-DBS 2: 50% reduction of left STN-DBS amplitude (voltage)
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
m/s | 0.941 (0.086) | -0.069 (0.048) | -0.016 (0.048)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; Bilateral (baseline) values are the average of the outcome measure data obtained during the 2 bilateral (baseline) conditions: 1) at enrollment before randomization and 2) after randomization. These average values are used to compare the changes associated with the 2 asymmetric conditions; Test type: Superiority; p = 0.163, Mixed Models Analysis — Holm-adjusted P-Value: 0.326 *Gait Velocity for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.749, Mixed Models Analysis — Holm-adjusted P-Value: 0.749 *Gait Velocity for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

2. Secondary Outcome: Change in Motor Function
Description: As measured by the MDS-UPDRS (Movement Disorders Society Unified Parkinson's Disease Rating Scale), which is a clinical and research tool to measure symptoms and signs of Parkinson's disease. It has 4 parts: I (non-motor experiences of daily living), II (motor experiences of daily living), III (motor exam) and IV (motor complications). The MDS-UPDRS has 60 items, scored from 0-4 each. The minimum score is 0 and the maximum score is 240.
  The MDS-UPDRS (motor) is Part III and measures motor signs. It has 28 items, scored from 0-4 each, so the minimum score is 0 and the maximum score is 112.
  The MDS-UPDRS (axial motor) is composed of items 3.1 to 3.3a and 3.9 to 3.13 of Part III of the MDS-UPDRS and measures axial motor signs. It has 8 items, scored from 0-4 each, so the minimum score is 0 and the maximum score is 32.
  In the MDS-UPDRS total, motor and axial motor sub-scales, lower scores indicate better symptoms/signs and higher scores indicate worse symptoms/signs, respectively.
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: Bilateral (baseline) values are the average of the outcome measure data obtained during the 2 bilateral (baseline) conditions: 1) at enrollment before randomization and 2) after randomization. These average values are used to compare the changes associated with the 2 asymmetric conditions.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
units on a scale
  MDS-UPDRS (total) | 1.032 (0.093) | 10.058 (4.491) | 1.277 (4.491)
  MDS-UPDRS (motor) | 1.080 (0.086) | 4.582 (2.147) | 1.636 (2.147)
  MDS-UPDRS (axial motor) | 0.947 (0.074) | -1.342 (0.823) | -2.453 (0.823)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; Bilateral (baseline) values are the average of the outcome measure data obtained during the 2 bilateral (baseline) conditions: 1) at enrollment before randomization and 2) after randomization. These average values are used to report the changes associated with the 2 asymmetric conditions; Test type: Superiority; p = 0.031, Mixed Models Analysis — Holm-adjusted P-Value: 0.155 *MDS-UPDRS (total) for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.778, Mixed Models Analysis — Holm-adjusted P-Value: 0.902 *MDS-UPDRS total for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 3: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.039, Mixed Models Analysis — Holm-adjusted P-Value: 0.157 *MDS-UPDRS (motor) for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 4: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.451, Mixed Models Analysis — Holm-adjusted P-Value: 0.902 *MDS-UPDRS (motor) for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 5: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.111, Mixed Models Analysis — Holm-adjusted P-Value: 0.333 *MDS-UPDRS (axial motor) for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 6: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.005, Mixed Models Analysis — Holm-adjusted P-Value: 0.030 *MDS-UPDRS (axial motor) for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

3. Secondary Outcome: Change in Axial Motor Function (1)
Description: As measured by the Mini-BESTest. The Mini-BESTest is a shorter version of the BESTest (Balance Evaluation Systems Test). It is a clinical and research tool to measure balance control. The Mini-BESTest has 14 items, scored from 0-2 each, so the minimum score is 0 and the maximum score is 28. Lower scores indicate worse balance control and higher scores indicate better balance control.
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
units on a scale | 0.967 (0.068) | -0.017 (0.828) | 1.557 (0.828)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.984, Mixed Models Analysis — Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.067, Mixed Models Analysis — Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

4. Secondary Outcome: Change in Axial Motor Function (2)
Description: As measured by the UPDRS-PIGD sub-scale. The UPDRS-PIGD is the Postural Instability Gait Dysfunction (PIGD) sub-scale of the Unified Parkinson's Disease Rating Scale (UPDRS). It is a clinical and research tool to measure PIGD. The UPDRS-PIGD has 5 items, scored from 0-4 each, so the minimum score is 0 and the maximum score is 20. Lower scores indicate better PIGD and higher scores indicate worse PIGD.
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
units on a scale | 0.909 (0.153) | -0.549 (0.704) | -1.414 (0.704)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.440, Mixed Models Analysis — Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.051, Mixed Models Analysis — Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

5. Secondary Outcome: Change in Axial Motor Function (3)
Description: As measured by the Freezing of Gait Questionnaire. The Freezing of Gait Questionnaire is a clinical and research tool to measure freezing of gait. It has 6 items, scored from 0-4 each, so the minimum score is 0 and the maximum score is 24. Lower scores indicate better and higher scores indicate worse freezing of gait, respectively.
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
units on a scale | 0.837 (0.088) | -0.056 (0.807) | -1.888 (0.807)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.945, Mixed Models Analysis — Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.024, Mixed Models Analysis — Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

6. Secondary Outcome: Change in Quantitative Gait Analysis (1)
Description: Changes in gait velocity in m/s as measured by a quantitative gait analysis system (Zeno walkway).
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: m/s
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
m/s | 0.814 (0.095) | -6.635 (3.910) | -1.254 (3.910)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.097, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Gait velocity for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.750, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Gait velocity for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

7. Secondary Outcome: Change in Quantitative Gait Analysis (2)
Description: Changes in step length in cm (mean, right, left) as measured by a quantitative gait analysis system (Zeno walkway).
  Step length difference = [right - left step length]
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
cm
  Step length (mean) | 0.975 (0.129) | -3.097 (1.990) | -3.191 (1.990)
  Step length (right) | 0.899 (0.156) | -2.867 (1.931) | -3.800 (1.931)
  Step length (left) | 1.015 (0.115) | -3.293 (2.252) | -3.493 (2.252)
  Step length difference | 0.731 (0.138) | 0.426 (1.088) | -0.307 (1.088)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.128, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Step length (mean) for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.117, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Step length (mean) for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 3: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.145, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Step length (right) for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 4: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.056, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Step length (right) for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 5: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.151, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Step length (left) for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 6: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.129, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Step length (left) for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 7: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.698, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Step length difference for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 8: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.779, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Step length difference for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

8. Secondary Outcome: Change in Quantitative Gait Analysis (3)
Description: Step length ratio = [right step length] / [left step length]
  Step length symmetry = ([right - left step length] / [right + left step length])
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
ratio
  Step length ratio | 1.214 (0.286) | -0.011 (0.071) | 0.002 (0.071)
  Step length symmetry | 0.934 (0.19) | 0.421 (2.36) | -0.420 (2.36)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.874, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Step length ratio for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.976, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Step length ratio for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 3: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.859, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Step length symmetry for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 4: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.860, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Step length symmetry for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

9. Secondary Outcome: Change in Quantitative Speech Analysis (1)
Description: Changes in pitch in Hertz (Hz) as measured by the Praat software.
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Hz
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
Hz
  Pitch (minimum) | 0.434 (0.242) | 16.864 (7.931) | 1.176 (7.931)
  Pitch (maximum) | 0.735 (0.071) | -146.413 (78.824) | -78.213 (78.824)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.040, Mixed Models Analysis — Holm-adjusted P-Value: 0.480 *Pitch (minimum) for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.883, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Pitch (minimum) for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 3: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.071, Mixed Models Analysis — Holm-adjusted P-Value: 0.781 *Pitch (maximum) for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 4: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.327, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Pitch (maximum) for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

10. Secondary Outcome: Change in Quantitative Speech Analysis (2)
Description: Changes in loudness in decibels (dB) as measured by the Praat software.
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: dB
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
dB
  Loudness (minimum) | 0.003 (0.048) | 0.549 (0.783) | 0.138 (0.783)
  Loudness (maximum) | 0.218 (0.083) | 0.619 (0.745) | -0.003 (0.745)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.487, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Loudness (minimum) for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.861, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Loudness (minimum) for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 3: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.411, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Loudness (maximum) for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 4: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.997, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Loudness (maximum) for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

11. Secondary Outcome: Change in Quantitative Speech Analysis (3)
Description: Changes in jitter measured in percentage by the Praat software. In this case, jitter is the percentage change in the stability of the frequency of speech tone (i.e. speech cycle-to-cycle frequency variation)
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change in speech tone freq.
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
percentage change in speech tone freq. | 1.263 (0.275) | 0.135 (0.155) | 0.063 (0.155)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.388, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Jitter for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.684, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Jitter for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

12. Secondary Outcome: Change in Quantitative Speech Analysis (4)
Description: Changes in shimmer measured in percentage by the Praat software. In this case, shimmer is the percentage change in the stability of the amplitude of speech tone (i.e. speech cycle-to-cycle amplitude variation)
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage change in speech tone amplit.
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
percentage change in speech tone amplit. | 0.630 (0.144) | -0.095 (0.498) | 0.185 (0.498)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.850, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Shimmer for Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.712, Mixed Models Analysis — Holm-adjusted P-Value: 1.00 *Shimmer for Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

13. Secondary Outcome: Change in Quality of Life
Description: As measured by the Total Score of the 39-item Parkinson's Disease Quality of Life Questionnaire (PDQ-39). The PDQ-39 is a clinical and research tool to measure quality of life in Parkinson's disease. It has 39 questions, which patients score as never (0% of the time), occasionally (25% of the time), sometimes (50% of the time), often (75% of the time) or always (100% of the time). The PDQ-39 Total Score or Summary Index is the average of the 39 questions, expressed. The minimum score is 0% (never) and the maximum score is 100% (always). Lower scores indicate better quality of life and higher scores indicate worse quality of life.
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 22 | 22 | 22
units on a scale | 0.792 (0.154) | 1.701 (2.506) | -3.148 (2.506)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.501, Mixed Models Analysis; Asymmetric STN-DBS 1 (right STN-DBS reduced) vs. Bilateral STN-DBS
Statistical Analysis 2: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 2; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.216, Mixed Models Analysis — Asymmetric STN-DBS 2 (left STN-DBS reduced) vs. Bilateral STN-DBS

14. Secondary Outcome: Change in Select Cognitive Tasks
Description: Left brain cognitive function: Hopkins Verbal Learning Test-Revised: Total recall trials 1-3 (0-36), delayed recall (0-12); Phonemic Verbal Fluency (0-no max); Semantic Verbal Fluency (Animal cue) (0-no max); Letter 1-back and 2-back working memory tasks (0-100%). Right brain cognitive function: Brief Visual Memory Test-Revised: Total recall trials 1-3 (0-36), delayed recall (0-12); Computerized landmark line bisection (-10 to 10); Spatial 1-back and 2-back working memory tasks (0-100%). Ranges in parentheses. Line bisection: closer to 0 is more accurate. For the rest: higher values are better
Time Frame: Baseline and 3 to 4 weeks after switching to each of the DBS conditions (Bilateral, Asymmetric 1, Asymmetric 2)
Population: Two patients could not complete cognitive tasks due to language barrier.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bilateral STN-DBS | Asymmetric STN-DBS 1 | Asymmetric STN-DBS 2
Number analyzed (Participants) | 20 | 20 | 20
units on a scale
  HopkinsVerbalLearningTest-Revised: RecallTrials1-3 | -0.30 (3.81) | 0.50 (3.90) | -0.85 (3.95)
  HopkinsVerbal LearningTest-Revised: Delayed Recall | -0.45 (2.04) | -0.75 (1.80) | -1.40 (2.48)
  Phonemic Verbal Fluency | 2.00 (7.05) | 2.70 (7.26) | 2.35 (8.38)
  Semantic Verbal Fluency (Animal cue) | 0.05 (6.16) | 0.50 (4.41) | 0.80 (3.79)
  Letter 1-Back Working Memory Task | 2.74 (16.46) | 4.44 (14.30) | 3.41 (15.68)
  Letter 2-Back Working Memory Task | 3.06 (17.35) | 0.95 (18.98) | 0.71 (16.83)
  Brief Visual Memory Test-Revised: RecallTrials 1-3 | 3.25 (4.55) | 3.45 (5.40) | 2.30 (4.40)
  Brief Visual Memory Test-Revised: Delayed Recall | 1.05 (2.39) | 1.55 (2.86) | 0.85 (2.87)
  Computerized landmark line bisection task | 0.05 (0.60) | 0.01 (0.77) | -0.02 (0.88)
  Spatial 1-Back Working Memory Task | -1.07 (17.19) | 0.31 (9.34) | -5.63 (14.65)
  Spatial 2-Back Working Memory Task | 0.16 (21.92) | -1.03 (24.01) | 1.67 (24.46)
Statistical Analysis 1: Comparison: Bilateral STN-DBS vs Asymmetric STN-DBS 1 vs Asymmetric STN-DBS 2; Test type: Superiority; p > 0.05, Friedman test — Non-adjusted P-Values were >0.05 and Holm-adjusted P-Values were 1.00 for all comparisons, except for the Hopkins Verbal Learning Test-Revised: Delayed Recall. For this test, the non-adjusted P-Value was 0.04 and the Holm-adjusted P-Value was 0.44; Using ranks for repeated measures (3 conditions)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 12-18 weeks (study duration per patient) plus at least 12 additional weeks for patients who opted for the open label phase after study completion.
Groups:
- Bilateral STN-DBS (Study Phase): Bilateral (baseline) STN-DBS settings (During the randomized, blinded phase)
- Asymmetric STN-DBS 1 (Study Phase): 50% reduction of right STN-DBS amplitude (voltage) (During the randomized, blinded phase)
- Asymmetric STN-DBS 2 (Study Phase): 50% reduction of left STN-DBS amplitude (voltage) (During the randomized, blinded phase)
- Asymmetric STN-DBS 1 (Open Label Phase): 50% reduction of right STN-DBS amplitude (voltage) (During the open label phase)
- Asymmetric STN-DBS 2 (Open Label Phase): 50% reduction of left STN-DBS amplitude (voltage) (During the open label phase)
Arm/Group | Bilateral STN-DBS (Study Phase) | Asymmetric STN-DBS 1 (Study Phase) | Asymmetric STN-DBS 2 (Study Phase) | Asymmetric STN-DBS 1 (Open Label Phase) | Asymmetric STN-DBS 2 (Open Label Phase)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/7 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22 | 0/22 | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 0/22 | 8/22 | 3/22 | 1/7 | 2/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bilateral STN-DBS (Study Phase) (N=22) | Asymmetric STN-DBS 1 (Study Phase) (N=22) | Asymmetric STN-DBS 2 (Study Phase) (N=22) | Asymmetric STN-DBS 1 (Open Label Phase) (N=7) | Asymmetric STN-DBS 2 (Open Label Phase) (N=10)
Treatment failure (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) — Patient did not tolerate this condition due to either 1) increase of 30% or more in the baseline MDS-UPDRS or 2) increase of less than 30% in the baseline MDS-UPDRS that did not respond to compensatory increase in the levodopa equivalent daily dose.
Increase in levodopa equivalent daily dose (Nervous system disorders) | 0 (0) | 5 (5) | 2 (2) | 0 (0) | 0 (0) — Patient required compensatory increase in levodopa equivalent daily dose in order to tolerate this condition (Increase of less than 30% in the baseline MDS-UPDRS that responded to compensatory increase in the levodopa equivalent daily dose)

LIMITATIONS AND CAVEATS:
There were no dropouts. The study phase of the trial concluded after the 22nd patient completed participation. As established by the sample size calculation, the originally planned enrollment of 27 patients was not necessary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-10-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT03462082/Prot_SAP_ICF_000.pdf